CLINICAL TRIAL: NCT00125658
Title: Mechanisms of Upper-Extremity Motor Recovery in Post-stroke Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B3964-R
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Cerebrovascular Accident
Keywords: biomechanics; Cerebrovascular Accident; electromyography; muscular weakness; recovery of function; reflex variability stroke; upper-extremity kinematics
MeSH Terms: conditions — Stroke; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): FTP: 30 sessions (90 minute sessions, 3 times per week, 10 weeks) followed by POWER: 30 sessions (90 minute sessions, 3 times per week, 10 weeks)
  Interventions: Other: Control
- Experimental (Experimental): POWER: 30 sessions (90 minute sessions, 3 times per week, 10 weeks) followed by FTP: 30 sessions (90 minute sessions, 3 times per week, 10 weeks)
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Control — Following an initial testing session, you will complete a 5 week no training period. At the end of this period you will then participate in a 20 week therapy program - 10 weeks of Functional Task Practice (FTP) followed by 10 weeks of Power training (dynamic resistance exercise). Each 10 week block has 30 therapy sessions for a total of 60 sessions, each lasting approximately 1-1/2 hours. Follow up evaluations will be scheduled at 6 months and 12 months after completion of the entire 20 week therapy program.
  Other Names: Order A
  Arms: Control
Other: Experimental — Following an initial testing session, you will complete a 5 week no training period. At the end of this period you will then participate in a 20 week therapy program - 10 weeks of Power training (dynamic resistance exercise) followed by 10 weeks of Functional Task Practice (FTP). Each 10 week block has 30 therapy sessions for a total of 60 sessions, each lasting approximately 1-1/2 hours. Follow up evaluations will be scheduled at 6 months and 12 months after completion of the entire 20 week therapy program.
  Other Names: Order B
  Arms: Experimental

SUMMARY:
The results of this study will provide sound, scientific evidence of physiologic mechanisms responsible for upper-extremity weakness; evidence of the processes involved in neuromuscular adaptation; and will elucidate the relationship between impairment and motor disability in post-stroke hemiparesis.

DETAILED DESCRIPTION:
This proposal extends the work accomplished in our initial study (project #B2405R, 'Effects of Strength Training on Upper-limb Function in Post-stroke Hemiparesis'). In the present study we will conduct a double-blind, randomized clinical trial of staged rehabilitation for the upper-extremity involving sequential delivery of functional therapy and high intensity resistance training. Therefore, this proposal directly compares the effects of functional and resistance training delivered individually. The researchers' previous work investigated a hybrid therapy of functional and resistance training against functional training alone. All subjects will participate in a 5 week run-in period of no treatment. This no-treatment block will afford multiple baseline measurements and, in addition, will provide information regarding the rate and magnitude of any spontaneous recovery without treatment. Following the second baseline measurement, all subjects will be randomized to upper-extremity rehabilitation in either: Order A - 10 weeks of functional task practice training (FTP) followed by 10 weeks of high-intensity resistance training (Power) or Order B - resistance training (Power) followed by FTP. Re-evaluation will occur following each block of treatment,and retention effects will be evaluated after 6 and 12 months with no additional treatment. Subjects will be evaluated with: outcome measures used broadly in Clinical Neurology and Rehabilitation, a battery of biomechanical performance measures including: strength, muscle activation, reflex modulation, and motor coordination, and with kinematics of free reaching movements. The researchers will investigate persons in the intermediate phase of recovery which they define as between 6 and 18 months post-stroke , having completed all inpatient and outpatient therapies, with remaining residual motor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cerebrovascular accident
* Single event
* Unilateral hemiplegia
* Between 6 months and 18 months post-event
* Impairment of upper-extremity function
* Ability to produce partial range of motion out of plane of gravity at shoulder, elbow, and wrist
* At least 10 degrees of wrist motion (any 10 degrees), and finger flexion/extension in 2 fingers
* Cognitive ability to follow 3-step commands

Exclusion Criteria:

* Unstable or uncontrolled blood pressure
* Uncontrolled seizures
* Flaccid hemiplegia
* Severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolynn Patten, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Corti M, McGuirk TE, Wu SS, Patten C. Differential effects of power training versus functional task practice on compensation and restoration of arm function after stroke. Neurorehabil Neural Repair. 2012 Sep;26(7):842-54. doi: 10.1177/1545968311433426. Epub 2012 Feb 22. PMID 22357633
- [Result] Phadke CP, Robertson CT, Condliffe EG, Patten C. Upper-extremity H-reflex measurement post-stroke: reliability and inter-limb differences. Clin Neurophysiol. 2012 Aug;123(8):1606-15. doi: 10.1016/j.clinph.2011.12.012. Epub 2012 Jan 23. PMID 22277759
- [Result] Phadke CP, Robertson CT, Patten C. Upper-extremity spinal reflex inhibition is reproducible and strongly related to grip force poststroke. Int J Neurosci. 2015 Jun;125(6):441-8. doi: 10.3109/00207454.2014.946990. Epub 2014 Sep 3. PMID 25135282

RESULTS

PARTICIPANT FLOW:
Groups:
- Order A (FTP Prior to Power): Participants randomized to Order A received 10 weeks of functional task practice (FTP) followed by 10 weeks of upper-extremity power training (Power).
- Order B (Power Prior to FTP): Participants randomized to Order B received 10 weeks of upper-extremity Power Training followed by 10 weeks of functional task practice (FTP).
Period: Overall Study
Arm/Group | Order A (FTP Prior to Power) | Order B (Power Prior to FTP)
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Order A: Participants randomized to Order A received 10 weeks of functional task practice (FTP) followed by 10 weeks of upper-extremity power training (Power).
  Single, unilateral stroke, >6 <26 months post-event.
- Order B: Participants randomized to Order B received 10 weeks of upper-extremity Power Training followed by 10 weeks of functional task practice (FTP).
  Single, unilateral stroke, >6 <26 months post-event.
- Total: Total of all reporting groups
Arm/Group | Order A | Order B | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (17.9) | 64.2 (9.8) | 59.8 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Trunk Displacement
Description: Distance (in cm) of trunk lean while performing reach-to-grasp. This information is obtained from kinematics/3D motion capture and is used to inform regarding compensatory use of the trunk as compared to active motion of the shoulder, elbow, wrist, and hand, during reach-to-grasp. Change scores are expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
centimeters
  Treatment effect (10 wks) | 3.79 (0.97) | -3.62 (1.81)
  Order effect (20 wks) | 0.66 (2.44) | -4.76 (2.82)
Statistical Analysis 1: Comparison: Order A vs Order B; Primary Comparison (i.e., FTP vs. POWER) Data are reported as change scores, between the end of treatment block 1(10 weeks) and baseline; thus, this analysis directly compares FTP vs. Power. A negative value represents improvement (i.e., reduced trunk displacement) while a positive value represents an increase in compensatory trunk movement; Test type: Superiority or Other; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Order A vs Order B; Order effect, testing OrderA (FTP before POWER) vs. OrderB (POWER before FTP). Change scores for trunk displacement at the end of both treatment blocks (20 weeks) relative to baseline (e.g., 20 weeks - baseline) were compared between OrderA and OrderB; Test type: Superiority or Other; p = .002, t-test, 2 sided

2. Primary Outcome: Change in Shoulder Flexion
Description: joint range of motion obtained using kinematics / motion capture. Change scores expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Order A: Participants randomized to Order A received 10 weeks of functional task practice (FTP) followed by 10 weeks of upper-extremity power training (Power).
- Order B: Participants randomized to Order B received 10 weeks of upper-extremity Power Training followed by 10 weeks of functional task practice (FTP).
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
degrees
  Treatment effect (10 wks) | -2.42 (10.44) | 11.88 (7.78)
  Order effect (20 wks) | -1.61 (10.81) | 10.37 (9.51)
Statistical Analysis 1: Comparison: Order A vs Order B; Tests effect of FTP vs. Power. The change in shoulder flexion range of motion was compared between baseline and the end of treatment Block 1 (i.e., 10 weeks); Test type: Superiority or Other; p = 0.13, t-test, 2 sided
Statistical Analysis 2: Comparison: Order A vs Order B; Test the effect of treatment order OrderA (FTP before POWER) vs. OrderB (POWER before FTP). The change in shoulder flexion range of motion was compared between the end of treatment (20 weeks) and baseline; Test type: Superiority or Other; p = 0.048, t-test, 2 sided

3. Primary Outcome: Change in Elbow Extension Range of Motion
Description: joint range of motion obtained using kinematics / motion capture. Change scores are expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
degrees
  Treatment effect (10 wks) | -8.83 (11.3) | 22.52 (20.3)
  Order effect (20 wks) | -5.62 (11.64) | 26.20 (30.58)
Statistical Analysis 1: Comparison: Order A vs Order B; Compares FTP vs POWER by comparing the change in elbow extension range of motion between the end of treatment block 1 (10 weeks) and baseline; Test type: Superiority or Other; p = .004, t-test, 2 sided
Statistical Analysis 2: Comparison: Order A vs Order B; Tests for the effect of treatment order OrderA (FTP before POWER) vs. OrderB (POWER before FTP) by comparing the change in elbow extension range of motion between the end of overall treatment (20 weeks) and baseline; Test type: Superiority or Other; p = 0.034, t-test, 2 sided

4. Secondary Outcome: Movement Speed
Description: peak velocity of movement (cm/s) during reach-to-grasp, obtained using kinematics/motion capture. Data are change scores expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
cm/s
  Treatment effect (10 wks) | 3.86 (4.21) | -2.67 (6.99)
  Order effect (20 wks) | 1.46 (7.20) | 7.15 (7.28)
Statistical Analysis 1: Comparison: Order A vs Order B; Tests for differences between FTP vs. POWER by comparing the change in movement speed between the end of treatment block 1 (10 weeks) and baseline; Test type: Superiority or Other; p = 0.056, t-test, 2 sided
Statistical Analysis 2: Comparison: Order A vs Order B; Tests for effect of treatment order (OrderA (FTP before POWER) vs. OrderB (POWER before FTP))by comparing the change in movement speed between the end of overall treatment (20 weeks) and baseline; Test type: Superiority or Other; p = .168, t-test, 2 sided

5. Primary Outcome: Upper-extremity Fugl-Meyer Motor Assessment
Description: The Fugl-Meyer Motor Assessment is a standardized scale used to measure the magnitude of motor impairment (severity) following stroke. There are separate sub-scales for the upper and lower extremities. Here we used the upper-extremity component; the full range of the scale is 0 - 66 points. Higher scores approaching 66 represent better, and lower scores approaching 0 worse, motor function. There is a significant ceiling effect with the FMA, thus a score of 66 points does not mean an individual with stroke has fully recovered. Data are change scores expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
units on a scale
  Treatment effect (10 wks) | 7.0 (9.1) | 6.7 (4.4)
  Order effect (20 wks) | 10.14 (4.34) | 9.00 (5.80)
Statistical Analysis 1: Comparison: Order A vs Order B; Tests the effects of FTP vs. POWER on motor impairment (UE FMA) by comparing the change in FMA between the end of treatment block 1 (10 weeks) and baseline; Test type: Superiority or Other; p = 0.564, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Order A vs Order B; Tests for an effect of treatment order (OrderA (FTP before POWER) vs. OrderB (POWER before FTP)) by comparing the change in UE FMA between the end of treatment (20 weeks) and baseline; Test type: Superiority or Other; p = 0.948, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Movement Accuracy (Reach Path Ratio, RPR)
Description: Measure is derived from kinematics/motion analysis. RPR = ratio of actual reach trajectory relative to an idealized straight line. Data are change scores, expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
ratio
  Treatment effect (10 wks) | -0.22 (1.70) | -1.82 (1.38)
  Order effect (20 wks) | -0.85 (1.72) | -1.59 (1.43)
Statistical Analysis 1: Comparison: Order A vs Order B; Tests for differences in FTP vs. POWER by comparing the change in RPR between the end of treatment block 1 (10 weeks) and baseline; Test type: Superiority or Other; p = 0.078, t-test, 2 sided
Statistical Analysis 2: Comparison: Order A vs Order B; Tests the effect of treatment order (Order A (FTP > POWER) vs. Order B (POWER > FTP)) by comparing the change in RPR between the end of overall treatment (20 weeks) and baseline; Test type: Superiority or Other; p = 0.4, t-test, 2 sided

7. Secondary Outcome: Movement Smoothness
Description: Movement smoothness is determined by assessing the number of sub movements (i.e., starts and stops) that can be identified during performance of a task. Here the task was reach-to-grasp. Sub movement are identified from kinematics/3D motion analysis. Sub-movements represent discontinuities or "jerky" movements. For example, skilled reaching is smooth and may reveal a single movement unit; in contrast, unskilled movements will reveal multiple movement units (i.e., starts and stops). As a performer practices and learns the movement, the number of sub movements is reduced. Sub movements can also present in persons with pathology. The unit of sub movements is whole numbers, or counts, of the sub movements. Data are change scores, expressed relative to baseline.
Time Frame: baseline, 10 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: sub movements
Arm/Group | Order A | Order B
Number analyzed (Participants) | 8 | 6
sub movements
  Treatment effect (10 wks) | 0.71 (4.43) | -2.79 (1.38)
  Order effect (20 wks) | -1.64 (10.81) | -2.71 (2.40)
Statistical Analysis 1: Comparison: Order A vs Order B; Tests for the effect of treatment (FTP vs. POWER) by comparing the change in movement smoothness between the end of treatment block 1 (10 weeks) and baseline; Test type: Superiority or Other; p = 0.085, t-test, 2 sided
Statistical Analysis 2: Comparison: Order A vs Order B; Tests for the effect of treatment order (OrderA (FTP before POWER) vs. OrderB (POWER before FTP)) by comparing the change in movement smoothness between the end of overall treatment (20 weeks) and baseline; Test type: Superiority or Other; p = 0.635, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Order A | Order B
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

LIMITATIONS AND CAVEATS:
This was a small clinical trial (total n = 14).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes